CLINICAL TRIAL: NCT06515626
Title: Clinical Study to Evaluate the Safety and Efficacy of Genetically Modified T Cells in the Treatment of Malignant Tumors
Brief Title: Genetically Modified T Cells Treating Malignant Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yi Zhang (Other)
Responsible Party: Sponsor-Investigator, Yi Zhang, M.D. &; Ph.D. Director, Biotherapy Center Co-Director, Division of Scientific Research Distinguished Professor, Cancer Center The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YiZhang
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Solid Tumor
Keywords: CAR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- subject (Experimental)
  Interventions: Biological: CAR-T cell reinfusion

INTERVENTIONS:
Biological: CAR-T cell reinfusion — Subjects were identified according to their benefit from the first treatment and target expression Whether to accept multiple returns; CAR-T cell reinfusion dose was 1~10×106 cells/kg, and the reinfusion dose could be adjusted according to the tolerance of the subjects Usually intravenous infusion, but also according to the need for local interventional treatment or injection treatment

SUMMARY:
To observe the safety, tolerability and initial effectiveness of gene modified T cell therapy in patients with malignant tumors in First Affiliated Hospital of Zhengzhou University, China.

DETAILED DESCRIPTION:
The study population included subjects with malignant tumors confirmed by histopathology or cytology, including: non-small cell lung cancer, esophageal squamous cell carcinoma, gastric cancer, colorectal cancer, liver cancer, pancreatic cancer, kidney cancer, cervical squamous cell carcinoma, ovarian cancer, breast cancer, melanoma, brain glioma, lymphoma, etc.

The study is aimed to observe the safety, tolerability and initial effectiveness of gene modified T cell therapy in patients with malignant tumors.To observe Progression-Free Survival (PFS) and Overall survival (OS) after the application of gene modified T cell therapy in patients with malignant tumors, and to evaluate the Disease Control Rate (Disease Control Rate). DCR, Clinical Benefit Rate (CBR), Quality of Life (QOL).And explore the diversity of T cell receptors and proportion of lymphocyte subsets in subjects treated with gene-modified T cell therapy for malignant tumors changes in distribution and count, immune cell function, and serum cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with malignant tumors confirmed by histopathology or cytology, including: non-small cell lung cancer, esophageal squamous cell carcinoma, gastric cancer, colorectal cancer, liver cancer, pancreatic cancer, kidney cancer, cervical squamous cell carcinoma, ovarian cancer, breast cancer, melanoma, and brain glia tumor, lymphoma, etc.;
2. Age: 18 ~ 75 years old; Gender: no limitation;
3. Have sufficient hematopoietic capacity: ANC >1500 cells /mm3, Blood plate count >50,000 cells /mm3, HGB >9.0g/dL, ALC >9 cells /mm3;
4. Adequate liver and kidney function: AST and ALT ≤2.5 ULN in patients without liver metastasis and ≤5 times in patients with liver metastasis. ULN; Bilirubin ≤1.5 ULN (excluding hyperbilirubinemia or hyperbilirubin of non-hepatic origin); Creatinine ≤2.0 ULN. Creatinine clearance and creatinine clearance hormone ≥40 mL/min;
5. PT/INR <1.5 ULN, and PTT/αPTT <1.5 ULN;
6. For desirable tumor tissues or tissue white tablets, positive expression of at least one of Mesothelin, NKG2D, HER2, CD276, CD19, BCMA and other antigens can be selected for clinical trials;
7. ECOG physical status score 0 ~ 2 points;
8. Expected survival >6 months;
9. Subject accepts voluntarily

Exclusion Criteria:

1. Received anti-PD1, anti-PD-L1 or anti-PD-L2 antibody therapy or other immunotherapy methods one month before treatment with immune cells in this study;
2. History of organ transplantation;
3. Pregnancy or lactation;
4. Positive for high baseline HBV DNA levels (≥2000 IU/ml), HIV antibodies (anti-HIV), hepatitis C virus antibodies (anti-HCV), or treponema pallidum antibodies;
5. There is active infection;
6. There are active brain metastases (except asymptomatic or stable brain metastases after treatment);
7. Combined with a second tumor; With the exception of patients with basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ, or papillary thyroid cancer who achieved complete response to the second tumor for more than 5 years and did not require treatment during the study period;
8. Severe autoimmune diseases such as ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, autoimmune vasculitis, or Wegener's granulomatosis require long-term (more than 2 months) systemic immunosuppressive therapy;
9. People with allergies;
10. NYHA heart failure grade ≥2 or hypertension can not be controlled after standard treatment, have a history of myocarditis or have a heart attack within one year;
11. Thrombotic diseases with active bleeding that require treatment;
12. Patients who are determined by the researcher to have a serious uncontrollable disease or other conditions that may affect the treatment in this study and are considered unsuitable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 36 months
  Progression-Free-Survival (PFS) is defined as admission to the group according to imaging specialists based on RECIST 1.1 review when disease progression or death from any cause was first recorded, whichever came first.

SECONDARY OUTCOMES:
OS | up to 36 months
  Overall survival (OS) is the time from enrollment to death from any cause
ORR | up to 36 months
  Objective response rate（ORR） refers to the proportion of subjects in the analysis population who achieved complete response (CR) or partial response (PR).
DOR | up to 36 months
  Duration of response (DOR). For subjects with confirmed CR or PR, duration of remission is the time from first recording to evidence of CR or PR until disease 2 progression (according to RECIST 1.1) or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Quality of life improvement | Baseline,The first day of each course (before dosing),up to 4weeks .
  EORTC QLQ C-30 survey

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, Study Chair — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Zhengzhou University First Affiliated Hospital, Zhengzhou, Henan, China